CLINICAL TRIAL: NCT02092636
Title: Ultrasound and Near Infrared Imaging for Breast Cancer Diagnosis and Neoadjuvant Chemotherapy Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Susan Tannenbaum, Associate Professor, UConn Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-194-6; R01EB002136 (NIH)
Record Dates: First submitted 2014-03-05; First posted 2014-03-20 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: Hybrid NIR/US imaging technique; NIR/US imaging; US imaging; US imaging technique
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NIR/US Diagnostic Group (Experimental): These patients will include women who have breast lumps/lesions visible by ultrasound and are prescribed follow up with an ultrasound-guided biopsy at the UCHC Cancer Center for evaluation and diagnosis of actual/suspected breast abnormalities.
  Interventions: Other: NIR/US Diagnostic Group
- NIR/US Neoadjuvant Chemotherapy Group (Experimental): These patients will include women who have breast lumps/lesions visible by ultrasound and have been diagnosed with breast cancers and will undergo neoadjuvant chemotherapy. These patients may be identified from the diagnostic group or after initial diagnosis. Patients will only be enrolled to one of the two groups.
  Interventions: Other: NIR/US Neoadjuvant Chemotherapy Group
- NIR/US Process Validation Group (Other): This group will contain data from about five women who did not have ultrasound visible lumps on the day of the planned biopsy. Data from the NIR/US scan will be used to validate instrument measurements.
  Interventions: Other: NIR/US Process Validation Group

INTERVENTIONS:
Other: NIR/US Diagnostic Group — Patients receiving an ultrasound-guided biopsy will participate in one study visit on the day of the biopsy. The NIR/US scan will be completed immediately prior to the biopsy procedure and takes about 5-10 minutes to perform.
  Arms: NIR/US Diagnostic Group
Other: NIR/US Neoadjuvant Chemotherapy Group — Patients may have the NIR/US scan performed at the time of their initial ultrasound-guided biopsy. In addition, patients in this group may also have NIR/US performed according the schedule in Table 1. The number of NIR/US study visits for these subjects will vary from 1-11 depending on the subject's treatment regimen. The expected duration of study participation for these patients is approximately 6 months.
  Arms: NIR/US Neoadjuvant Chemotherapy Group
Other: NIR/US Process Validation Group — Patients who present with visible lumps at initial ultrasound but do not have ultrasound visible lumps on the day of the biopsy procedure will not require a biopsy. NIR/US scan will be performed. Data from the NIR/US scan will be used to validate instrument measurements.
  Arms: NIR/US Process Validation Group

SUMMARY:
An imaging method has been developed that uses near infrared light as an adjunct to ultrasound for better diagnosis and for monitoring tumor response. This study will use a new, non-invasive way to evaluate breast lumps using a low power light source & ultrasound to see if breast lumps are benign or cancerous. This study will also evaluate if this new technique might be useful in assessing response to chemotherapy.

DETAILED DESCRIPTION:
The investigators propose to validate the utility of the investigators novel hybrid imaging technique for accurate diagnosis of breast lesions, and for assessing chemotherapy response of cancer treatment and predicting treatment efficacy. The investigators unique hybrid technique is implemented by simultaneously deploying near infrared (NIR) optical sensors and a commercial ultrasound (US) transducer mounted on a hand-held probe, and utilizing co-registered lesion structure information provided by ultrasound to improve the inverse optical tomography reconstruction. As a result, the optical tomography assisted with US has overcome problems associated with intense light scattering and has provided reliable tumor angiogenesis distributions. Initial results with a group of 200 biopsied patients have shown that early stage invasive cancers present two-fold greater total hemoglobin concentration on average than fibroadenomas and other benign lesions. Initial results of advanced cancers have shown that the angiogenesis distribution is highly distorted and heterogeneous, and the distorted distributions correlate with histological microvessel density counts and can be used to assess chemotherapy response.

Objective of this study is to validate the investigators initial results that NIR light guided by ultrasound can improve breast cancer diagnosis and monitor chemotherapy response.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older who have breast lumps or abnormalities (actual or suspected) are eligible for the study.
* Women and members of all races and ethnic groups are eligible for this study.
* Diagnostic Group: These patients will include women who have breast lumps/lesions visible by ultrasound and are prescribed follow up with an ultrasound-guided biopsy at the UCHC Cancer Center for evaluation and diagnosis of actual/suspected breast abnormalities.
* Neoadjuvant Chemotherapy Group: These patients will include women who have breast lumps/lesions visible by ultrasound and have been diagnosed with breast cancers and will undergo neoadjuvant chemotherapy. These patients may be identified from the diagnostic group or after initial diagnosis. Patients will only be enrolled to one of the two groups.
* Process Validation Group: This group will contain data from about five women who did not have ultrasound visible lumps on the day of the planned biopsy. Data from the NIR/US scan will be used to validate instrument measurements.

Exclusion Criteria:

* All Subjects who fail to meet the inclusion criteria are ineligible for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Hemoglobin concentration | 5 years
  The deoxygenated/oxygenated hemoglobin and total hemoglobin concentration are the measured imaging parameters and biopsy results will be used as the 'gold' standard to compare imaging findings. Hemoglobin concentration is measured in micromolar/liter.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Tannenbaum, MD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided.

REFERENCES:
- [Derived] Zhu Q, Tannenbaum S, Kurtzman SH, DeFusco P, Ricci A Jr, Vavadi H, Zhou F, Xu C, Merkulov A, Hegde P, Kane M, Wang L, Sabbath K. Identifying an early treatment window for predicting breast cancer response to neoadjuvant chemotherapy using immunohistopathology and hemoglobin parameters. Breast Cancer Res. 2018 Jun 14;20(1):56. doi: 10.1186/s13058-018-0975-1. PMID 29898762